CLINICAL TRIAL: NCT01029808
Title: Bleeding Symptoms of Carriers of Hemophilia A and B
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Anna Olsson, MD, Sahlgrenska University Hospital
Other Study IDs: VGAO002
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Hemophilia
Keywords: carriers of hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To collect and analyze data on female carriers of severe and moderate hemophilia A and B.

ELIGIBILITY:
Inclusion Criteria:

* Female carriers of hemophilia A and B.

Exclusion Criteria:

* Pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Carriers of severe and moderate hemophilia A and B
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Bleeding tendency in carriers of severe and moderate haemophilia compared to a control group. | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Baghaei, MD PhD, Study Chair
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Sweden

REFERENCES:
- [Result] Olsson A, Hellgren M, Berntorp E, Ljung R, Baghaei F. Clotting factor level is not a good predictor of bleeding in carriers of haemophilia A and B. Blood Coagul Fibrinolysis. 2014 Jul;25(5):471-5. doi: 10.1097/MBC.0000000000000083. PMID 24509327
- [Result] Olsson A, Hellgren M, Berntorp E, Baghaei F. Association between bleeding tendency and health-related quality of life in carriers of moderate and severe haemophilia. Haemophilia. 2015 Nov;21(6):742-6. doi: 10.1111/hae.12796. Epub 2015 Sep 8. PMID 26346645